CLINICAL TRIAL: NCT02187627
Title: Evaluation of [11C]RO6924963, [11C]RO6931643, and [18F]RO6958948 as Tracers for Tau Imaging With Positron Emission Tomography in Healthy Control Subjects and Subjects With Alzheimer's Disease
Brief Title: Evaluation of [11C]RO6924963, [11C]RO6931643, and [18F]RO6958948 as Tracers for Positron Emission Tomography (PET) Imaging of Tau in Healthy and Alzheimer's Disease (AD) Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: BP29409
Record Dates: First submitted 2014-06-17; First posted 2014-07-11 (Estimated); Last update posted 2019-01-02 (Actual); Status verified 2018-12

CONDITIONS: Alzheimer's Disease, Healthy Volunteer
MeSH Terms: conditions — Alzheimer Disease

ARMS (3):
- Part 1: Tracer Selection (Experimental): Participants will receive a single dose of one tracer on one occasion and a single dose of a different tracer after 7 to 14 days and will be followed for 7 to 14 days for safety. At the end of Part 1, one tracer with the best performance will be selected for further study in Part 2.
  Interventions: Drug: [11C]RO6924963; Drug: [11C]RO6931643; Drug: [18F]RO6958948
- Part 2A: Test-Retest (Experimental): Participants will receive a single dose of selected tracer from Part 1 on one occasion and then same tracer will be administered after 6 weeks. Participants will be followed for 7 to 14 days after last PET tracer administration for safety.
  Interventions: Drug: [11C]RO6924963; Drug: [11C]RO6931643; Drug: [18F]RO6958948
- Part 2B: Dosimetry (Experimental): Participants will receive a single dose of selected tracer from Part 1 and will be followed for 7 to 14 days for evaluation of radiation dosimetry.
  Interventions: Drug: [11C]RO6924963; Drug: [11C]RO6931643; Drug: [18F]RO6958948

INTERVENTIONS:
Drug: [11C]RO6924963 — Radiolabeled low molecular weight compound, administered as single intravenous injection. The mass dose of [11C]RO6924963 injected will be </=10 micrograms (mcg), injection volume </=20 milliliters (mL). Target injected activity for [11C]RO6924963 will be 370-740 megabecquerel (MBq) [10-20 millicurie (mCi)].
Drug: [11C]RO6931643 — Radiolabeled low molecular weight compound, administered as single intravenous injection. The mass dose of [11C]RO6931643 injected will be </=10 mcg, injection volume </=20 mL. Target injected activity for [11C]RO6931643 will be 370-740 MBq (10-20 mCi).
Drug: [18F]RO6958948 — Radiolabeled low molecular weight compound, administered as single intravenous injection. The mass dose of [18F]RO6958948 injected will be </=10 mcg, injection volume </=20 mL. Target injected activity for [18F]RO6958948 will be 185-370 MBq (5-10 mCi). The final activity of [18F] RO6958948 will be adjusted up to 10 mCi per scan to allow sufficient counts by end of 200 minutes post radiotracer injection.

SUMMARY:
This study is designed to obtain basic information on three PET imaging tracers developed to detect tau pathology in the brain. In this study, healthy control participants and participants with AD will be studied. Information collected will include brain and plasma kinetics, tissue distribution (in the brain), radiation dosimetry, and test-retest variability of the signal in the brain. The study will consist of Part 1, Part 2A, and Part 2B. During Part 1, imaging data will be assessed on an ongoing basis and based on data, one tracer will be prioritized over the other two tracers. The tracer selected will be further investigated in Part 2A and Part 2B.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria for All Participants

* Agreement to use highly effective contraception measures
* If participants are on any concomitant medication, the indication and dosage of these medicines should be stable for at least 4 weeks prior to study start with the expectation that no relevant changes in use or dose will occur throughout the study
* Body mass index (BMI) between 18 and 32 kilograms per square meter (kg/m^2)
* Weight less than or equal to (</=) 300 pounds (lb)

Inclusion Criteria for Healthy Control Participants

* Healthy "young" control participants aged 25-40 years or healthy "elderly" control participants aged greater than or equal to (>/=) 50 years
* Normal cognitive function, including a normal Mini Mental State Examination (MMSE) score as judged by the investigator
* Healthy control participants who participate in Part 2B: must be less than (<) 195 centimeter (cm) (6 feet, 5 inches) tall in order to accommodate the whole body scanning

Inclusion Criteria for Participants with a Diagnosis of Probable AD

* Diagnosis of probable AD, according to the National Institute of Neurological and Communicative Disorders and Stroke/Alzheimer's Disease and Related Disorders Association criteria
* Participants aged >/= 50 years
* A study partner able to accompany the participant to all visits and answer questions about the participant
* MMSE score between 16 and 26, inclusive

Exclusion Criteria:

Exclusion Criteria for All Participants

* History or presence of a neurological diagnosis other than AD that may influence the outcome or analysis of the scan results; examples include but are not limited to stroke, traumatic brain injury, space occupying lesions, non-Alzheimer's tauopathies, and Parkinson's disease
* Participants with a medical history that includes known autosomal dominant AD mutations in amyloid precursor protein (APP) or presenilin (PS1, PS2) or mutations in genes that cause other types of autosomal dominant familial dementia
* History or presence of any clinically relevant hematological, hepatic, respiratory, cardiovascular, renal, metabolic, endocrine, or central nervous system disease or other medical conditions that are not well controlled, may put the participant at risk, could interfere with the objectives of the study, or make the participant unsuitable for participation in the study for any other reason in the opinion of the principal investigator
* Clinically relevant pathological findings in physical examination, electrocardiogram, or laboratory values at the screening assessment that could interfere with the objectives of the study
* Known history of clinically significant infectious disease including acquired immunodeficiency syndrome (AIDS) or serological indication of acute/chronic hepatitis B or C or human immunodeficiency virus infection
* Pregnancy or lactation
* Unsuitable veins for repeated venipuncture
* Current symptoms of allergy and/or severe allergy to drugs in medical history
* Alcohol consumption that averages >3 drinks daily or regular smoker (>10 cigarettes, >3 pipefuls, or >3 cigars per day)
* Coffee (or tea) consumption >10 cups per day or methylxanthine-containing drinks >1.5 liters per day (L/day)
* Have received an investigational medication within the last 3 months or 5 times (x) the elimination half-life, whichever is longer, prior to Day 1 (i.e., enrollment)

Exclusion Criteria Related to Trial Procedures

* Presence of pacemakers; aneurysm clips; artificial heart valves; ear implants; foreign metal objects in the eyes, skin, or body, or any other circumstance (e.g. claustrophobia) that would contraindicate a magnetic resonance imaging (MRI) scan
* For participants of Part 1 and Part 2A, any contraindications to arterial cannulation

Exclusion Criterion for Participants with Probable Alzheimer's Disease

* Has received treatment that targeted amyloid-beta or tau within the last 24 months

Min Age: 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2014-08-31 (Actual); Primary Completion 2016-02-29 (Actual); Study Completion 2016-02-29 (Actual)

PRIMARY OUTCOMES:
Part 1: Standard Uptake Value (SUV), as Assessed by Tau PET Brain Scan | Day 1 up to Day 14
Part 1: Standard Uptake Value Ratio (SUVR), as Assessed by Tau PET Brain Scan | Day 1 up to Day 14
Part 1: SUV, as Assessed by Tau PET Scan of Whole Body | Day 1 up to Day 14
Part 1: SUVR, as Assessed by Tau PET Scan of Whole Body | Day 1 up to Day 14
Mean Residence Times for Each Organ, as Assessed by Tau PET Scan of Whole Body | Day 1 up to Day 14
Part 1: Distribution Volume (VT), as Assessed by Tau PET Brain Scan | Day 1 up to Day 14

SECONDARY OUTCOMES:
Part 2A: Absolute Percentage Difference Between Test and Retest of SUVR | Days 1, 28
Part 2A: Absolute Percentage Difference Between Test and Retest of VT | Days 1, 28
Part 2B: Effective dose (ED), as Assessed by Whole Body PET Scan | From the time of tracer injection on Day 1 up to 120 minutes post injection
Part 2A: Absolute Percentage Difference Between Test and Retest of SUV | Days 1, 28
Percentage of Participants With Adverse Events (AEs) | Part 1: Day 1 up to Day 28, Part 2a: Day 1 up to Day 42, Part 2b: Day 1 up to Day 15

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (2):
- United States (2):
  - Parexel International; Harbor Hospital Center, Baltimore, Maryland
  - Johns Hopkins Universtiy; Radiology Dept, Baltimore, Maryland